CLINICAL TRIAL: NCT06043492
Title: Recovery Following Different Endurance Training Protocols in Middle- and Long-Distance Runners
Brief Title: Recovery Following Acute Endurance Training
Acronym: ETRec
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Thessaly (Other)
Responsible Party: Principal Investigator, Chariklia K. Deli, Assistant Professor, University of Thessaly
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Screening
Other Study IDs: Endurance Training - Recovery
Record Dates: First submitted 2023-09-17; First posted 2023-09-21 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: High Intensity Interval Training; Continuous Running; Control Condition
MeSH Terms: interventions — High-Intensity Interval Training

STUDY DESIGN:
Intervention Model Description: The same participants will participate in three different conditions
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- High Intensity Interval Training (Experimental): The participants will perform an acute bout of high intensity interval training
  Interventions: Other: High Intensity Interval Training
- Coninuous Running (Experimental): The participants will perform an acute bout of continuous running
  Interventions: Other: Coninuous Running
- Control Trial (Other): The participants will not perform any endurance exercise protocol
  Interventions: Other: Control Trial

INTERVENTIONS:
Other: High Intensity Interval Training — 10 x 2 min running at vVO2max, interspersed by 2 min recovery at 40% VO2max
  Arms: High Intensity Interval Training
Other: Coninuous Running — 40 min continuous running at lactate threshold
  Arms: Coninuous Running
Other: Control Trial — The participants will perform only the baseline and post acute-training evaluations, without performing exercise
  Arms: Control Trial

SUMMARY:
Aerobic capacity is critical for many athletes, especially for endurance athletes. Althgough several training methods are implemented by coaches to improve endurance performance, recovery following acute endurance training is not adequately studied. However, such information is crucial for coaches to effectively design the most favorable training program, to avoid muscle injuries and overtraining, and ultimately to improve performance of their athletes. This study aims to examine the acute effect of different continuous and HIIT training protocols on indices of metabolism, EIMD, neuromuscular fatigue and performance in middle- and long-distance runners.

DETAILED DESCRIPTION:
Aerobic capacity is critical for many athletes, especially for endurance athletes. Endurance training leads to cardiopulmonary and musculoskeletal adaptations, which in turn lead to improvement of endurance performance. Several training methods have been established for the improvement of aerobic capacity and performance, including long distance and low speed training, and high intensity interval training (HIIT). Training methods are used depending on the kind of endurance that aim to improve, and the specific characteristics and energy demands of the event. Especially regarding middle- and long-distance runners, the energy comes mainly from the oxidative system, however, the contribution of the glycolytic pathway is equally important. Thus, improvement mainly of the low-intensity endurance, but also high-intensity endurance is important for these athletes. Additionally, both continuous endurance and HIIT are effective training methods for improving cardiorespiratory and metabolic function, and athletic performance, while evidence also exists in favor of HIIT being more effective. Thus both training methods are used by coaches to improve aerobic capacity and performance of their athletes.

Coaches should be careful regarding the frequency of HIIT training during a microcycle, to provide adequate recovery between training sessions to avoid muscle injuries and overtraining. Existing evidence suggests that endurance exercise (continuous or HIIT) may result in exercise-induced muscle damage (EIMD), inflammatory responses, oxidative stress, and performance deterioration, yet, the timeframe of recovery of physiological and biochemical indices following different endurance training protocols has not been adequately studied. However, such information is crucial for coaches to effectively design the most favorable training program for their athletes.

This study aims to examine the acute effect of different continuous and HIIT training protocols on indices of metabolism, EIMD, neuromuscular fatigue and performance in middle- and long-distance runners.

According to a preliminary power analysis (a probability error of 0.05, and a statistical power of 80%), a sample size of 8 subjects per group was considered appropriate in order to detect statistically meaningful changes between groups. Thus, 10 men and female middle- and long-distance runners, will participate in the study.

The study will be performed in a randomized, cross over, repeated measures design. During their first 1st and 2nd visit, all participants will sign an informed consent form after they will be informed about all the benefits and risks of the study and they will fill in and sign a medical history questionnaire. Fasting blood samples will be collected in order to estimate muscle damage concentration markers. Participants will be instructed by a dietitian how to record a 7-days diet recalls to ensure that they do not consume to greater extent nutrients that may affect EIMD and fatigue (e.g. antioxidants, amino acids, etc.) and to ensure that the energy intake during the trials will be the same. Assessment of body mass and body height, body composition, and aerobic capacity (VO2max), will be performed. Using a photocells system, countermovement jump will be performed to assess jump height, and 30 sec Bosco test to assess mean jump height, peak power, mean power, and fatigue index. The peak concentric, eccentric and isometric isokinetic torque of the knee flexors and extensors, in both limbs will be evaluated on an isokinetic dynamometer at 60°/sec. Maximal voluntary isometric contraction (MVIC) of the knee extensors at 65o in both limbs, as well as the fatigue rate during MVIC through the percent drop of peak torque between the first and the last three seconds of a 10-sec MVIC, will also be evaluated. Afterwards, participants will be randomly assigned into, and perform one of the three different conditions of the study design: a) Continuous running (CT) for 40 min at lactic threshold, b) High intensity interval training (HIIT): 10x2min running at vVO2max with active recovery at 40% της VO2max (interval:recovery 1:1) with a load of 10% of body weight (BW), and c) control condition, no training (measurements only). The training protocols will be matched for mean power and total duration (Tschakert and Hofmann 2013). Prior and immediately after each experimental trial, delayed onset of muscle soreness (DOMS) in the knee flexors (KF) and extensors (KE) of both limbs, as well as blood lactate will be assessed. Additionally, DOMS of KF and KE, peak concentric, eccentric and isometric isokinetic torque, CMJ height, as well as mean jump height, peak power, mean power, and fatigue index during a 30 sec Bosco test, will be assessed 24h, 48h and 72h after the end of the trial. MVIC of the knee extensors of both limbs, as well as the fatigue rate during MVIC will also be assessed at 1h, 2h and 3h, as well as 24h, 48h, and 72h after the end of the trial. Creatine kinase will be assessed at 24h, 48h, and 72h after the end of the trial. The exact above procedures will be repeated by the participants during the remaining two experimental trials. A 2-weeks wash-out period will be implemented between trials.

ELIGIBILITY:
Inclusion Criteria:

* Middle- and long-distance runners
* Absence of musculoskeletal injuries (≥ 6 months)
* No use of drugs or ergogenic supplements (≥ 1 month)
* Absense from eccentric exercise (≥ 3 days)
* No alcohol or ergogenic drinks consumption before each training protocol

Exclusion Criteria:

* Musculoskeletal injury (< 6 months)
* Use of drugs or ergogenic supplements (< 1 month)
* Participation in eccentric exercise (< 3 days)
* Alcohol or ergogenic drinks consumption before the training protocol

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2023-09-30 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2023-12-15 (Actual)

PRIMARY OUTCOMES:
Changes in Creatine kinase (CK) | Baseline (pre), 24 hours post-, 48 hours post-, 72 hours post-trial
  CK will be measured in plasma using a Clinical Chemistry Analyzer with commercially available kits.
Changes in DOMS | Baseline (pre), post-, 24 hours post-, 48 hours post-, 72 hours post-trial
  DOMS of knee extensors and knee flexors of both lower extremities will be measured during palpation of the muscle belly and the distal region after performing three repetitions of a full squat.
Changes in blood lactate | Baseline (pre), 4 minutes post-trial
  Lactate will be measured in capillary blood with a hand-portable analyzer.
Changes in squat jump height | Baseline (pre), 24 hours post-, 48 hours post-, 72 hours post-trial
  Squat jump height will be measured with a photocells system.
Changes in mean jump height during a 30 sec Bosco test | Baseline (pre), 24 hours post-, 48 hours post-, 72 hours post-trial
  Mean jump height will be measured with a photocells system.
Changes in peak power during a 30 sec Bosco test | Baseline (pre), 24 hours post-, 48 hours post-, 72 hours post-trial
  Peak power will be measured with a photocells system.
Changes in mean power during a 30 sec Bosco test | Baseline (pre), 24 hours post-, 48 hours post-, 72 hours post-trial
  Mean power will be measured with a photocells system.
Changes in fatigue rate during a 30 sec Bosco test | Baseline (pre), 24 hours post-, 48 hours post-, 72 hours post-trial
  Fatigue rate will be estimated through the persent drop in mean jump height between the first 5 jumps and the last 5 jumps.
Changes in maximal voluntary isometric contraction (MVIC) | Baseline (pre), 1 hour post-, 2 hours post-, 3 hours post-, 24 hours post-, 48 hours post-, 72 hours post-trial
  MVIC of the knee extensors and knee flexors will be measured on an isokinetic dynamometer.
Changes in peak concentric torque | Baseline (pre), 24 hours post-, 48 hours post-, 72 hours post-trial
  Concentric torque of the knee extensors and knee flexors will be measured on an isokinetic dynamometer.
Changes in peak eccentric torque | Baseline (pre), 24 hours post-, 48 hours post-, 72 hours post-trial
  Eccentric torque of the knee extensors and knee flexors will be measured on an isokinetic dynamometer.

SECONDARY OUTCOMES:
Body weight | Baseline
  Body weight will be measured on a beam balance with stadiometer.
Body height | Baseline
  Body height will be measured on a beam balance with stadiometer.
Body mass index (BMI) | Baseline
  BMI will be calculated from the ratio of body mass/ body height squared.
Body fat | Baseline
  Body fat will be measured by using Dual-emission X-ray absorptiometry.
Lean body mass | Baseline
  Lean body mass will be measured by using Dual-emission X-ray absorptiometry.
Dietary intake | Baseline
  Dietary intake will be assessed using 7-day diet recalls.
Maximal oxygen consumption (VO2max) | Baseline
  VO2max will be measured by open circuit spirometry via breath by breath method during a graded treadmill running protocol.

CONTACTS AND LOCATIONS:
Overall Officials: Chariklia K Deli, PhD, Principal Investigator — University of Thessaly
Locations (1):
- Department of Physical Education and Sport Science, Uninersity of Thessaly, Trikala, Thessaly, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Barnes KR, Kilding AE. Strategies to improve running economy. Sports Med. 2015 Jan;45(1):37-56. doi: 10.1007/s40279-014-0246-y. PMID 25164465
- [Background] Brandao LHA, Chagas TPN, Vasconcelos ABS, de Oliveira VC, Fortes LS, de Almeida MB, Mendes Netto RS, Del-Vecchio FB, Neto EP, Chaves LMS, Jimenez-Pavon D, Da Silva-Grigoletto ME. Physiological and Performance Impacts After Field Supramaximal High-Intensity Interval Training With Different Work-Recovery Duration. Front Physiol. 2020 Oct 8;11:1075. doi: 10.3389/fphys.2020.01075. eCollection 2020. PMID 33162893
- [Background] Cipryan L. IL-6, Antioxidant Capacity and Muscle Damage Markers Following High-Intensity Interval Training Protocols. J Hum Kinet. 2017 Mar 15;56:139-148. doi: 10.1515/hukin-2017-0031. eCollection 2017 Feb. PMID 28469752
- [Background] Esfarjani F, Laursen PB. Manipulating high-intensity interval training: effects on VO2max, the lactate threshold and 3000 m running performance in moderately trained males. J Sci Med Sport. 2007 Feb;10(1):27-35. doi: 10.1016/j.jsams.2006.05.014. Epub 2006 Jul 28. PMID 16876479
- [Background] Hottenrott K, Ludyga S, Schulze S. Effects of high intensity training and continuous endurance training on aerobic capacity and body composition in recreationally active runners. J Sports Sci Med. 2012 Sep 1;11(3):483-8. eCollection 2012. PMID 24149357
- [Background] Martinez-Ferran M, Cuadrado-Penafiel V, Sanchez-Andreo JM, Villar-Lucas M, Castellanos-Montealegre M, Rubio-Martin A, Romero-Morales C, Casla-Barrio S, Pareja-Galeano H. Effects of Acute Vitamin C plus Vitamin E Supplementation on Exercise-Induced Muscle Damage in Runners: A Double-Blind Randomized Controlled Trial. Nutrients. 2022 Nov 3;14(21):4635. doi: 10.3390/nu14214635. PMID 36364898